CLINICAL TRIAL: NCT01309282
Title: Portuguese Observational Re-Treatment Study of MabThera (PORTSMAB) - A Two-centre Observational Study in Sero-positive Rheumatoid Arthritis (RA) Patients Who Are Non-responders or Intolerant to a Single Tumor Necrosis Factor (TNF) Inhibitor
Brief Title: An Observational Study of MabThera/Rituxan (Rituximab) in Patients With Sero-Positive Rheumatoid Arthritis Who Are Non-Responders or Intolerant to a Single TNF-Inhibitor (PORTSMAB)
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML22935
Record Dates: First submitted 2011-03-03; First posted 2011-03-07 (Estimated); Results first posted 2016-04-21 (Estimated); Last update posted 2016-08-12 (Estimated); Status verified 2016-08

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Rituximab: Sero-positive [Rheumatoid Factor (RF) and/or anti-Cyclic Citrullinated Peptide (CCP+)] rheumatoid arthritis (RA) patients, who had initiated therapy with Rituximab (MabThera) following lack of response or intolerance to a single tumour necrosis factor (TNF)-inhibitor will be included in this arm

SUMMARY:
This observational study will assess the long-term efficacy and safety of MabThera/Rituxan in routine clinical practice in patients with sero-positive rheumatoid arthritis who are non-responders or intolerant to a single tumour necrosis factor (TNF) inhibitor. Data will be collected from each patient over 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Rheumatoid arthritis positive for rheumatoid factor and/or anti-CCP
* Non-responder or intolerant to single TNF-inhibitor therapy
* Initiating treatment with MabThera/Rituxan

Exclusion Criteria:

* Contra-indications to MabThera/Rituxan therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with sero-positive rheumatoid arthritis starting treatment with MabThera/Rituxan following lack of response or intolerance to single TNF-inhibitor
Sampling Method: Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2010-07; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Lisbon, Portugal

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 9 participants were enrolled in one center from Portugal between 01 Jul 2010 and 30 Jun 2011. The first participant's screening visit was on 01 Jul 2010 and the last participant's last visit was on 19 Aug 2013. Although it was initially planned to involve two centers, it was only possible to involve a single center.
Groups:
- Rituximab: Participants with sero-positive [Rheumatoid Factor (RF) and/or anti-Cyclic Citrullinated Peptide (CCP+)] rheumatoid arthritis (RA), who had commenced therapy with rituximab (MabThera) following lack of response or intolerance to a single tumor necrosis factor (TNF)-inhibitor were included in this arm.
Period: Overall Study
Arm/Group | Rituximab
Started | 9
Completed | 8
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least one dose of study drug, whether prematurely withdrawn from the study or not and who complied with the criteria for inclusion.
Groups:
- Rituximab: Participants with sero-positive (RF and/or CCP+) RA, who had commenced therapy with rituximab following lack of response or intolerance to a single TNF-inhibitor, were included in this arm.
Arm/Group | Rituximab
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.78 (14.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 1

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Disease-activity Score 28-Erythrocyte Sedimentation Rate at Month 24
Description: The disease-activity score 28 (DAS28) score is a measure of validated instrument for the assessment of the overall severity of RA disease activity calculated using the tender joint count (TJC), swollen joint count (SJC), patient's global assessment of disease activity, and erythrocyte sedimentation rate (ESR) for a total possible score of 2 to 10. Higher values indicate higher disease activity. A negative change from baseline indicates improvement.
Time Frame: Baseline (Day 0) and Month 24
Population: The analysis was conducted with all the participants who complied with the inclusion and exclusion criteria, thus defining full analysis set (n=9). However, data is presented only for those participants who completed Month 24 visit (n=8).
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Rituximab
Number analyzed (Participants) | 8
Scores on a scale | -2.31 (0.88)
Statistical Analysis 1: Comparison: Rituximab; Test type: Superiority or Other; p = 0.0078, Wilcoxon signed rank test

2. Secondary Outcome: Mean Change From Baseline in TJC at Month 24
Description: A tender joint count (TJC) is the most specific clinical method to quantify abnormalities in participants with RA. It is associated with the level of pain. Twenty-eight joints were assessed for tenderness. Joints were classified as tender (1)/not tender (0) giving a total possible TJC score of 0 to 28. A negative change from baseline indicates improvement.
Time Frame: Baseline (Day 0) and Month 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Tender joints
Arm/Group | Rituximab
Number analyzed (Participants) | 8
Tender joints | -7.5 (6.48)
Statistical Analysis 1: Comparison: Rituximab; Test type: Superiority or Other; p = 0.0078, Wilcoxon signed rank test

3. Secondary Outcome: Mean Change From Baseline in SJC at Month 24
Description: A swollen joint count (SJC) is the most specific clinical method to quantify abnormalities in participants with RA. It reflects the amount of inflamed synovial tissue. Twenty-eight joints were assessed for swelling. Joints were classified as swollen (1)/ not swollen (0) giving a total possible SJC score of 0 to 28. A negative change from baseline indicates improvement.
Time Frame: Baseline (Day 0) and Month 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Swollen joints
Arm/Group | Rituximab
Number analyzed (Participants) | 8
Swollen joints | -4.13 (2.30)
Statistical Analysis 1: Comparison: Rituximab; Test type: Superiority or Other; p = 0.01403, Wilcoxon signed rank test

4. Secondary Outcome: Mean Change From Baseline in ESR at Month 24
Description: The ESR is an acute phase reactant and a measure of inflammation. A negative change from baseline indicates improvement.
Time Frame: Baseline (Day 0) and Month 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Millimeter (mm)/hour
Arm/Group | Rituximab
Number analyzed (Participants) | 8
Millimeter (mm)/hour | -28.50 (29.66)
Statistical Analysis 1: Comparison: Rituximab; Test type: Superiority or Other; p = 0.0355, Wilcoxon signed rank test

5. Secondary Outcome: Mean Change From Baseline in C-reactive Protein at Month 24
Description: The C-reactive protein is an inflammation marker. High levels of this protein indicate inflammation in diseases such as RA. A negative change from baseline indicates improvement.
Time Frame: Baseline (Day 0) and Month 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Milligrams/liter
Arm/Group | Rituximab
Number analyzed (Participants) | 8
Milligrams/liter | -8.11 (24.42)
Statistical Analysis 1: Comparison: Rituximab; Test type: Superiority or Other; p = 0.5469, Wilcoxon signed rank test

6. Secondary Outcome: Mean Change From Baseline in Physician's Global Assessment of Disease Activity At Month 24
Description: The Physician's Global Assessment of disease activity was assessed using a Visual Analogue Scale (VAS). The left-hand extreme of the line equals 0 mm, and is described as "no disease activity" (symptom-free and no arthritis symptoms) and the right-hand extreme equals 100 mm, as "maximum disease activity" (maximum arthritis disease activity).Change from Baseline = score at observation minus score at Baseline. An increase in score from Baseline represents disease progression and/or joint worsening, no change represents halting of disease progression, and a decrease represents improvement.
Time Frame: Baseline (Day 0) and Month 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Rituximab
Number analyzed (Participants) | 8
Scores on a scale | -34.29 (13.94)
Statistical Analysis 1: Comparison: Rituximab; Test type: Superiority or Other; p = 0.0225, Wilcoxon signed rank test

7. Secondary Outcome: Mean Change From Baseline in Patient's Global Assessment of Disease Activity at Month 24
Description: The Patient's Global Assessment of disease activity was assessed using VAS. The left-hand extreme of the line equals 0 mm, and is described as "no disease activity" (symptom-free and no arthritis symptoms) and the right-hand extreme equals 100 mm, as "maximum disease activity" (maximum arthritis disease activity).Change from Baseline = score at observation minus score at Baseline. An increase in score from Baseline represents disease progression and/or joint worsening, no change represents halting of disease progression, and a decrease represents improvement.
Time Frame: Baseline (Day 0) and Month 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Rituximab
Number analyzed (Participants) | 8
Scores on a scale | -28.50 (20.71)
Statistical Analysis 1: Comparison: Rituximab; Test type: Superiority or Other; p = 0.0225, Wilcoxon signed rank test

8. Secondary Outcome: Mean Change From Baseline in Severity of Pain at Month 24
Description: The patient's assessment of pain was performed using a 100 mm VAS ranging from no pain (0) to unbearable pain (100). The distance in mm from the left edge of the scale was measured. A negative change from Baseline score indicates improvement in pain intensity.
Time Frame: Baseline (Day 0) and Month 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Rituximab
Number analyzed (Participants) | 8
Scores on a scale | -23.15 (30.48)
Statistical Analysis 1: Comparison: Rituximab; Test type: Superiority or Other; p = 0.0904, Wilcoxon signed rank test

9. Secondary Outcome: Mean Change Form Baseline in Functional Capacity at Month 24
Description: The functional capacity was analyzed using Health Assessment Questionnaire-Disability Index (HAQ-DI). It is a 20-question instrument that assesses the degree of difficulty a person has in accomplishing tasks in 8 domains (dressing, arising, eating, walking, hygiene, reaching, gripping and activities of daily living). Responses in each domain are scored from 0 to 3 (0=no difficulty; 1=some difficulty; 2=much difficulty; 3=unable to do). Overall score was computed as sum of domain scores and divided by the number of domains. A total possible score ranged from 0 (best) to 3 (worst).
Time Frame: Baseline (Day 0) and Month 24
Population: The analysis was conducted with all the participants who complied with the inclusion and exclusion criteria, thus defining full analysis set (n=9). However, the results are presented only for the participants with available data and who completed Month 24 visit (n=7).
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Rituximab
Number analyzed (Participants) | 7
Scores on a scale | -0.27 (0.59)
Statistical Analysis 1: Comparison: Rituximab; Test type: Superiority or Other; p = 0.2969, Wilcoxon signed rank test

10. Secondary Outcome: Reason for Change From First TNF-inhibitor Therapy to Rituximab
Description: Adverse event, primary and secondary insufficient responses and monoclonal gammopathy were the reasons for starting rituximab therapy.
Time Frame: At Screening
Population: The analysis was conducted with all 9 participants who complied with the inclusion and exclusion criteria, thus defining the full analysis set.
Measure: Number; unit: Participants
Arm/Group | Rituximab
Number analyzed (Participants) | 9
Participants
  Adverse event - esophageal candidiasis | 1
  Insufficient Response: Primary | 1
  Insufficient Response: Secondary | 6
  Monoclonal gammopathy | 1

11. Secondary Outcome: Number of Participants on Each Pattern of Re-treatment
Description: There are two patterns of re-treatment, namely treat-to-target and according to the clinic.
  Treat-to-target: a new cycle every 6 months if not in remission, with the participant receiving no new course of treatment as long as he is in remission.
  On demand (according to clinic): a new cycle when, in an assessment performed at least 16 weeks after the last treatment cycle, the participant shows moderate or high disease activity [DAS28 > 3.2 or difference in DAS28 (ΔDAS28) > 0.6]
Time Frame: Up to Month 24
Population: as for outcome 10
Measure: Number; unit: Participants
Arm/Group | Rituximab
Number analyzed (Participants) | 9
Participants
  Treat-to-target | 9
  On demand (according to clinic) | 0

12. Secondary Outcome: Number of Participants With Incidence of Infusion Reactions or Injection Site Reactions
Description: An infusion reaction or injection site reaction is an event that occurs after infusion or injection which may include hypersensitivity reactions or anaphylactic reactions.
Time Frame: At Months 6, 12 and 24
Population: Safety population was used for the analysis which included all participants who received at least one dose of study drug, whether prematurely withdrawn from the study or not and who complied with the criteria for inclusion.
Measure: Number; unit: Participants
Arm/Group | Rituximab
Number analyzed (Participants) | 9
Participants
  Month 6 | 0
  Month 12 | 0
  Month 24 | 1

13. Secondary Outcome: Number of Participants With Incidence of Infectious Events
Description: Follow-up of the infectious events was done after Month 6 visit, Month 12 visit and Month 24 visit.
Time Frame: At Months 6, 12 and 24
Population: as for outcome 12
Measure: Number; unit: Participants
Arm/Group | Rituximab
Number analyzed (Participants) | 9
Participants
  Month 6 | 0
  Month 12 | 2
  Month 24 | 0

14. Secondary Outcome: Number of Participants Who Experienced Any Adverse Events or Serious Adverse Events
Description: An Adverse Events (AE) is any untoward medical occurrence in a participant or clinical investigation subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. A Serious Adverse Events (SAE) is any untoward medical occurrence that at any dose results in death, are life threatening, requires hospitalization or prolongation of hospitalization or results in disability/incapacity, and congenital anomaly/birth defect
Time Frame: Up to Month 24
Population: as for outcome 12
Measure: Number; unit: Participants
Arm/Group | Rituximab
Number analyzed (Participants) | 9
Participants
  Any AEs | 5
  Any SAEs | 0

ADVERSE EVENTS:
Time Frame: Up to Month 24
Description: All AEs and SAEs were collected for Safety population which included all participants who received at least one dose of study drug, whether prematurely withdrawn from the study or not and who complied with the criteria for inclusion.
Arm/Group | Rituximab
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 5/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab (N=9)
Odynophagia (Gastrointestinal disorders) | 1
Idiosyncratic drug reaction (General disorders) | 1
Cutaneous lupus erythrematosus (Immune system disorders) | 1
Lower respiratory tract infection (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 1
Neutrophil count decreased (Investigations) | 1
White blood cell count decreased (Investigations) | 1
Left ankle fracture (Musculoskeletal and connective tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.